CLINICAL TRIAL: NCT05550259
Title: Evaluation of an Oxygenation and Ventilation Support Protocol for the PREvenTion of EXTubation Failure: a Stepped Wedge Cluster Randomized Trial
Brief Title: Ventilation Support for the PREvenTion of EXTubation Failure
Acronym: PRETEEXT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3480
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Extubation Failure

STUDY DESIGN:
Intervention Model Description: A stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control period (No Intervention): the control period corresponds to usual care of centers
- protocolized period (Experimental): the protocolized period corresponds to a protocolized use of HFNO or NIV after extubation
  Interventions: Procedure: protocolized postextubation support

INTERVENTIONS:
Procedure: protocolized postextubation support — The intervention corresponds to a protocolized use of HFNO or NIV after extubation in accordance with the risk of extubation failure: a) 24H HFNO in patient at low risk of extubation failure b) 48H NIV+/-HFNO in patients at high risk of extubation failure
  Arms: protocolized period

SUMMARY:
Reintubation after failed extubation would be associated with increased mortality. Therefore, extubation failure remains a major concern in ICU. Few randomized controlled studies have assessed the benefit for a systematic respiratory support (noninvasive ventilation or high flow nasal cannula) applied at the time of extubation to reduce reintubation rates in patients at high and low risk for reintubation. In addition, these studies reported discordant results. Therefore, there are some concerns regarding effectiveness and systematic uptake of a respiratory support after extubation into usual practice.

DETAILED DESCRIPTION:
The aim of this trial is to determine whether a protocolized postextubation respiratory support including High-flow Nasal Oxygen (HFNO) and Noninvasive Ventilation (NIV) could reduce the rate of reintubation in comparison with usual practice. Therefore, all consecutively eligible patients for the study, will be assigned to a protocol arm in accordance with the randomized period

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Intubated more than 24 hours in the ICU
* Ready for a scheduled extubation then extubated

Exclusion Criteria:

* Contraindication to HFNO or NIV
* Underlying chronic neuromuscular disease
* Unplanned extubation (accidental or self-extubation)
* With a do-not-reintubate order at time of extubation
* Tracheotomia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Rate of reintubation | 7 days following extubation
  Reintubation following extubation